CLINICAL TRIAL: NCT05857215
Title: A Phase 1, Double-blind, Single and Multiple-Dose Study of Safety, Tolerability and Pharmacokinetics of Amilo-5MER in Healthy Volunteers
Brief Title: A First-in-Human Study of Single and Multiple Doses of Amilo-5MER in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galmed Pharmaceuticals Ltd (Industry)
Collaborators: Quotient Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Amilo-5MER-002
Record Dates: First submitted 2023-04-25; First posted 2023-05-12 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-04

CONDITIONS: Inflammatory Disease

STUDY DESIGN:
Intervention Model Description: Part 1 of the study was a double-blind, randomised, placebo-controlled assessment of single subcutaneous (SC) ascending doses of amilo-5MER in healthy young adult male subjects. Subjects were enrolled sequentially into 1 of up to 5 cohorts, each containing 8 subjects
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Subjects were assigned to a treatment using a computer-generated randomization schedule.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- A- amilo-5MER solution for subcutaneous administration or matching placebo- 10 mg (Experimental): Amilo-5MER solution for subcutaneous administration or matching placebo at a dose of 10 mg
  Interventions: Drug: amilo-5MER
- B- amilo-5MER solution for subcutaneous administration or matching placebo- 30 mg (Experimental): Amilo-5MER solution for subcutaneous administration or matching placebo at a dose of 30 mg
  Interventions: Drug: amilo-5MER
- C- amilo-5MER solution for subcutaneous administration or matching placebo- 90 mg (Experimental): Amilo-5MER solution for subcutaneous administration or matching placebo at a dose of 90 mg
  Interventions: Drug: amilo-5MER
- D- amilo-5MER solution for subcutaneous administration or matching placebo- 180 mg (Experimental): Amilo-5MER solution for subcutaneous administration or matching placebo at a dose of 180 mg
  Interventions: Drug: amilo-5MER
- E- amilo-5MER solution for subcutaneous administration or matching placebo- 360mg (Experimental): Amilo-5MER solution for subcutaneous administration or matching placebo at a dose of 360 mg
  Interventions: Drug: amilo-5MER

INTERVENTIONS:
Drug: amilo-5MER — amilo-5MER is a 5 amino acid synthetic peptide MTADV (Methionine, Threonine, Alanine, Aspartic acid, Valine).
  Other Names: Synthetic peptide consisting of 5 amino acids

SUMMARY:
This is a three-part, single Centre, double-blind, randomized, placebo-controlled first-in-human study of single ascending doses (SADs, Part 1) and multiple doses (Part 2) of amilo-5MER in healthy young adult male subjects and a single dose cohort in healthy elderly male and female subjects (Part 3)

DETAILED DESCRIPTION:
This is a three-part, single Centre, double-blind, randomized, placebo-controlled first-in-human study of single ascending doses (SADs, Part 1) and multiple doses (Part 2) of amilo-5MER in healthy young adult male subjects and a single dose cohort in healthy elderly male and female subjects (Part 3).

The study aim is to assess and characterize the safety and tolerability of single and multiple doses of amilo-5MER in healthy young adult subjects and single doses in healthy elderly subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males (all parts) or healthy females (Part 3 only).
2. Aged 18 to 45 years (Parts 1 and 2) or aged 65 to 80 years (Part 3) inclusive at the time of signing informed consent.
3. Body mass index (BMI) of 19.0 to 31.0 kg/m2, with a body weight <95 kg, as measured at screening.
4. Willing and able to communicate and participate in the whole study.
5. Provided a written informed consent.
6. Agreed to adhere to the contraception requirements

Exclusion Criteria:

1. Subjects who had received any IMP in a clinical research study within the 90 days prior to Day 1.
2. Subjects who were, or were immediate family members of, a study site or sponsor employee.
3. Subjects who had previously been administered IMP in this study. Subjects who took part in Part 1 were not permitted to take part in Part 2.
4. Evidence of recent SARS-CoV-2 symptomatic infection within the last 3 months. Subjects who had asymptomatic, incidental, positive polymerase chain reaction (PCR) findings could have been included if tested more than 30 days prior to screening and test negative at screening.
5. History of any drug or alcohol abuse in the past 2 years.
6. Regular alcohol consumption in males >21 units per week and females (Part 3 only) >14 units per week (1 unit = ½ pint beer, or a 25 mL shot of 40% spirit, 1.5 to 2 units = 125 mL glass of wine, depending on type).
7. A confirmed positive alcohol breath test at screening or admission.
8. Current smokers and those who had smoked within the last 6 months. A confirmed breath carbon monoxide (CO) reading of greater than 10 ppm at screening or admission.
9. Current users of e-cigarettes and nicotine replacement products and those who had used these products within the last 6 months.
10. Females of childbearing potential including those who were pregnant or lactating (all female subjects must have had a negative highly sensitive urine and serum pregnancy test). A woman was considered of childbearing potential unless she was permanently sterile (hysterectomy, bilateral salpingectomy, and bilateral oophorectomy) or was postmenopausal (had no menses for 12 months without an alternative medical cause and a serum follicle stimulating hormone [FSH] concentration ≥30 IU/L) at screening and admission visit (Part 3 only).
11. Male subjects who had pregnant or lactating partners.
12. Subjects who did not have suitable veins for multiple venepunctures/cannulation as assessed by the investigator at screening.
13. Clinically significant abnormal clinical chemistry, haematology or urinalysis as judged by the investigator (laboratory parameters are listed in Appendix 1 of protocol [Appendix 16.1.1.1]).
14. Confirmed positive drugs of abuse test result (drugs of abuse tests are listed in Appendix 1 of protocol [Appendix 16.1.1.1]) at screening or admission.
15. Positive hepatitis B surface antigen (HBsAg), hepatitis C virus antibody (HCV Ab) or human immunodeficiency virus (HIV) antibody results.
16. Evidence of renal impairment at screening, as indicated by an estimated creatinine clearance (CLcr) of <80 mL/min (Parts 1 and 2) or <60 mL/min (Part 3) using the Cockcroft-Gault equation at screening.
17. History of clinically significant cardiovascular, renal, hepatic, dermatological, chronic respiratory or gastrointestinal disease, neurological or psychiatric disorder, as judged by the investigator.
18. Clinically significant abnormalities on electrocardiogram (ECG) (e.g. prolonged QTc, prolonged PR interval).
19. Serious adverse reaction or serious hypersensitivity to any drug or the formulation excipients.
20. Presence or history of clinically significant allergy requiring treatment, as judged by the investigator. Hay fever was allowed unless it was active.
21. Donation of blood or plasma within the previous 3 months or loss of greater than 400 mL of blood.
22. Had received blood or plasma derivatives in the 3 months preceding dosing.
23. Adherence (for whatever reason) to an abnormal diet during the 4 weeks prior to the study, or subjects with recent significant change in body weight.
24. Subjects who were taking, or had taken, any prescribed or over-the-counter drug (other than up to 2 g of paracetamol per day until 24 h prior to dosing and hormone replacement therapy [HRT]) or herbal remedies or dietary supplements (including bran) in the 14 days before IMP administration.
25. Subjects with tattoos or scars on the abdomen which could have interfered with injection site assessments, as determined by the investigator at screening.
26. Failure to satisfy the investigator of fitness to participate for any other reason.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-07-01 (Actual); Study Completion 2021-07-01 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability of amilo-5ER | 10 days
  Assess and characterize the number of participants with clinically significant changes in safety assessments, including adverse events, physical examination findings, vital signs, clinical laboratory assessments, and urinalysis.

SECONDARY OUTCOMES:
PK- Area under the concentration-time curve (AUC) | 10 days
  Investigate the plasma Area under the concentration-time curve (AUC) of single and multiple doses of amilo-5MER
PK- Time of maximum observed concentration (Tmax) | 10 days
  Investigate the plasma Time of maximum observed concentration (Tmax) of single and multiple doses of amilo-5MER
PK- Maximum observed concentration (Cmax) | 10 days
  Investigate the plasma Maximum observed concentration (Cmax) of single and multiple doses of amilo-5MER
PK- Total body clearance (CL/F) | 10 days
  Investigate the Total body clearance (CL/F) of single and multiple doses of amilo-5MER

CONTACTS AND LOCATIONS:
Overall Officials: John Posner, PhD, FRCP, Study Director — Pharmaceutical medicine consultant
Locations (1):
- Quotient Sciences, Mere Way, Ruddington, Nottingham, NG11 6JS, UK, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No
Data collected for exploration only.